CLINICAL TRIAL: NCT00568269
Title: Randomized Multicentre Study Comparing TEP With Lichtenstein Repair for Primary Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Stig and Ragna Gorthon Foundation (Unknown); Tyco Healthcare Group (Industry)
Responsible Party: Arne Eklund, MD, Centre for Clinical Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMIL II; Ups 144-96
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Inguinal Hernia
Keywords: Recurrence rate after inguinal hernia repair on primary inguinal herina.
MeSH Terms: conditions — Hernia, Inguinal

ARMS (2):
- Lichtenstein (Active Comparator)
  Interventions: Procedure: Open repair
- TEP (Experimental)
  Interventions: Procedure: Laparoscopic repair

INTERVENTIONS:
Procedure: Open repair — Open repair is according to the Lichtenstein technique
  Arms: Lichtenstein
Procedure: Laparoscopic repair — The TEP (Totally ExtraPeritoneal patch) repair is used as the laparoscopic repair
  Arms: TEP

SUMMARY:
The purpose of this study was to compare the recurrence rate after TEP (laparoscopic method) and Lichtenstein (open method) repair on primary inguinal hernia.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 30-70 years referred to hospital with a primary inguinal hernia.

Exclusion Criteria:

* Recurrent hernia
* Scrotal or bilateral hernia
* Previous lower abdominal surgery
* Unable to participate in follow up
* ASA more than 3
* Bleeding diathesis.

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1513 (Actual)
Dates: Start 1996-11; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | 5 years

SECONDARY OUTCOMES:
Operative complications, postoperative recovery and chronic pain at 5 years. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Arne S Eklund, MD, Principal Investigator — Centre for Clinical Research
Locations (1):
- Centre for Clinical Research, Central hospital, entrance 29, Västerås, Sweden

REFERENCES:
- [Result] Eklund A, Rudberg C, Smedberg S, Enander LK, Leijonmarck CE, Osterberg J, Montgomery A. Short-term results of a randomized clinical trial comparing Lichtenstein open repair with totally extraperitoneal laparoscopic inguinal hernia repair. Br J Surg. 2006 Sep;93(9):1060-8. doi: 10.1002/bjs.5405. PMID 16862612
- [Derived] Eklund A, Montgomery A, Bergkvist L, Rudberg C; Swedish Multicentre Trial of Inguinal Hernia Repair by Laparoscopy (SMIL) study group. Chronic pain 5 years after randomized comparison of laparoscopic and Lichtenstein inguinal hernia repair. Br J Surg. 2010 Apr;97(4):600-8. doi: 10.1002/bjs.6904. PMID 20186889